CLINICAL TRIAL: NCT02525861
Title: A Phase 3/4 Study to Evaluate the Safety, Immunogenicity, and Effects on the Alpha1-Proteinase Inhibitor (A1PI) Levels in Epithelial Lining Fluid Following Glassia Therapy in A1PI-Deficient Subjects
Brief Title: GLASSIA Safety, Immunogenicity, and Bronchoalveolar Lavage Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 471101
Record Dates: First submitted 2015-08-14; First posted 2015-08-18 (Estimated); Results first posted 2021-10-14 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-07

CONDITIONS: Alpha1-antitrypsin Deficiency
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency | interventions — alpha 1-Antitrypsin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort I: GLASSIA (High-end) (Experimental): Participants will receive weekly IV infusions of GLASSIA (lot with particle loads representing the high end within) at 60 milligrams per kilogram (mg/kg) BW active A1PI protein administered at a rate of 0.2 milliliters per kilogram of body weight per minute (ml/kg/min) for 25 weeks (25 planned infusions) via an IV administration.
  Interventions: Biological: GLASSIA
- Cohort II: GLASSIA (Low-end) (Experimental): Participants will receive weekly IV infusions of GLASSIA (lot with particle loads representing the low end within the normal range) at 60 mg/kg BW active A1PI protein administered at a rate of 0.2 ml/kg/min for 25 weeks (25 planned infusions) via an IV administration.
  Interventions: Biological: GLASSIA

INTERVENTIONS:
Biological: GLASSIA — Participants will receive weekly IV infusions of GLASSIA at 60 mg/kg BW active A1PI protein administered at a rate of 0.2 mL/kg/min for 25 weeks (25 planned infusions) via an IV administration.
  Other Names: Alpha1-Proteinase Inhibitor; A1PI

SUMMARY:
The purpose of the study is 2-fold: (1) to evaluate the safety and potential immunogenicity of GLASSIA following intravenous (IV) administration via in-line filtration; and (2) to assess the effects of GLASSIA augmentation therapy on the levels of A1PI and various biomarkers in the epithelial lining fluid (ELF) following intravenous (IV) administration at a dosage of 60 milligrams per kilogram (mg/kg) Body weight (BW)/week active alpha1-proteinase inhibitor (A1PI) protein for 25 weeks in participants with emphysema due to congenital A1PI deficiency.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants meeting the following age criteria:

   1. For participants who will undergo bronchoscopy/ bronchoalveolar lavage (BAL) procedures: 18 to 75 years of age at the time of screening.
   2. For participants who will be waived from undergoing bronchoscopy/BAL procedures: 18 years of age or older at the time of screening.
2. Documented Alpha1-Proteinase Inhibitor (A1PI) genotype of Pi*Z/Z, Pi*Z/Null, Pi*Malton/Z, Pi*Null/Null, or other "at-risk" allelic combinations such as SZ (excluding MS and MZ without the presence of another allowable at-risk genotype) and an endogenous A1PI plasma levels of less than or equal to (< or =)11 micrometer (μM) (< or = 0.572 milligrams per milliliter [mg/mL]).
3. Screening levels of endogenous plasma (antigenic) A1PI of < or =11 μM may be collected at any time during the screening period for treatment-naive participants, or following a 4 week minimum wash-out from previous augmentation therapy in treatment-experienced participants.
4. Participants must have at least one of the following: clinical diagnosis of emphysema, evidence of emphysema on computerized tomography (CT) scan of the chest, and/or evidence of airway obstruction which is not completely reversed with bronchodilator treatment at the time of screening.
5. If the participant is being treated with any respiratory medications including inhaled bronchodilators, inhaled anticholinergics, inhaled corticosteroids, or low-dose systemic corticosteroids (prednisone < or =10 milligram per day (mg/day) or its equivalent), the doses of the participant's medications have remained unchanged for at least 14 days prior to screening.
6. The participant is a nonsmoker or has ceased smoking for a minimum of 13 weeks prior to screening (serum cotinine level at screening within normal range of a nonsmoker) and agrees to refrain from smoking throughout the course of the study. Participants with a positive cotinine test due to nicotine replacement therapy (example [eg], patches, chewing gum), vapor cigarettes, or snuff are eligible.
7. If female of childbearing potential, the participant presents with a negative pregnancy test at screening and agrees to employ adequate birth control measures for the duration of the study.
8. The participant is willing and able to comply with the requirements of the protocol.
9. The participant must have pulmonary function at the time of screening meeting both of the following:

   1. Post-bronchodilator forced expiratory volume in 1 second (FEV1) greater than or equal to (> or =) 50 percentage (%) of predicted.
   2. If FEV1 is >80% predicted, then FEV1/forced vital capacity (FVC) must be <0.7. *Note: Inclusion criterion #1a, #9a and #9b are not applicable to participants who are not required to undergo the bronchoscopy/BAL procedures.

Exclusion Criteria:

1. The participant is experiencing or has a history of clinically significant pulmonary disease (other than chronic obstructive pulmonary disease (COPD), emphysema, chronic bronchitis, mild bronchiectasis, and stable asthma).
2. The participant is experiencing or has a history of chronic severe cor pulmonale (resting mean pulmonary artery pressure > or =40 millimeters) of mercury [mm Hg]).
3. The participant routinely produces more than 1 tablespoon of sputum per day.
4. The participant has a history of frequent pulmonary exacerbations (greater than 2 moderate or severe exacerbations within 52 weeks prior to screening.
5. The participant is experiencing a pulmonary exacerbation at the time of screening (participant may be rescreened 4 weeks after the clinical resolution of an exacerbation).
6. The participant has clinically significant abnormalities (other than emphysema, chronic bronchitis, or mild bronchiectasis) detected on chest X-ray or CT scan at the time of screening (past records obtained within 52 weeks prior to screening may be used, if available).
7. The participant has clinically significant abnormalities detected on a 12-lead electrocardiogram (ECG) performed at the time of screening (past records obtained within 26 weeks prior to screening may be used, if available).
8. The participant has clinically significant congestive heart failure with New York Heart Association (NYHA) Class III/IV symptoms.
9. The participant is experiencing an active malignancy or has a history of malignancy within 5 years prior to screening, with the exception of the following: adequately treated basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, or stable prostate cancer not requiring treatment.
10. The participant has a history of lung or other organ transplant, is currently on a transplant list, or has undergone major lung surgery.
11. The participant is receiving long-term around-the-clock oxygen (O2) supplementation. (The following are allowed: short-term use of oxygen supplementation [eg, for the management of acute COPD exacerbation], O2 supplementation required during night time only, and supplemental O2 with continuous positive airway pressure [CPAP] or bi-level positive airway pressure [BiPAP]).
12. Known history of hypersensitivity following infusions of human blood or blood components.
13. Immunoglobulin A (IgA) deficiency (<8 milligram per deciliter (mg/dL) at screening).
14. Abnormal clinical laboratory results obtained at the time of screening meeting any of the following criteria:

    1. Serum alanine aminotransferase (ALT) >3.0 times upper limit of normal (ULN)
    2. Serum total bilirubin >2.0 times ULN
    3. >2+proteinuria on urine dipstick analysis
    4. Serum creatinine >2.0 times ULN
    5. Absolute neutrophil count (ANC) <1500 cells per cubic millimeter (cells/mm^3)
    6. Hemoglobin (Hgb) <9.0 gram per deciliter (g/dL)
    7. Platelet count <100,000/cubic millimeter (mm^3)
15. Ongoing active infection with hepatitis A virus (HAV), hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV) Type 1 or 2 infection at the time of screening.
16. The participant has any clinically significant medical, psychiatric, or cognitive illness, or any other uncontrolled medical condition (eg, unstable angina, transient ischemic attack) that, in the opinion of the investigator, would impede the participant's ability to comply with the study procedures, pose increased risk to the participant's safety, or confound the interpretation of study results.
17. The participant has participated in another clinical study involving an IP or investigational device within 30 days prior to enrollment or is scheduled to participate in another clinical study involving an IP or device during the course of this study.
18. The participant is a family member or employee of the investigator.
19. If female, the participant is nursing at the time of screening.

    Note: Exclusion criteria #20, #21, #22, #23, and #24 are not applicable to participants who are not required to undergo the bronchoscopy/BAL procedures.
20. The participant has contraindication(s) to bronchoscopy such as recent myocardial infarction, unstable angina, other cardiopulmonary instability, tracheal obstruction or stenosis, moderate to severe hypoxemia or any degree of hypercapnia, unstable asthma, Stage 4 or 5 chronic kidney disease, pulmonary hypertension, severe hemorrhagic diathesis, and cervical C1/C2 arthritis.
21. The participant has had lung surgery which may interfere with bronchoscopy.
22. Known history of allergic/hypersensitivity reactions to medications used during and for perioperative care associated with the bronchoscopy/BAL procedures, such as local anesthetics, sedatives, pain control medications.
23. The participant is receiving or requires long-term (>4 weeks) immunosuppressive therapy, such as systemic corticosteroids at doses greater than 10 mg/day of prednisone (or its equivalent), mycophenolate mofetil, azathioprine, cyclophosphamide, and rituximab.
24. If a participant is receiving anticoagulant or anti-platelet therapy (such as warfarin and clopidogrel), the participant is unwilling to or unable to safely discontinue anticoagulant or anti-platelet therapy within 7 days prior to until at least 24 hours after the BAL procedures. An exception is low-dose aspirin alone which is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-03-08 (Actual); Primary Completion 2020-07-29 (Actual); Study Completion 2020-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (18):
- United States (17):
  - Arizona Board of Regents, University of Arizona, Tucson, Arizona
  - UCLA Medical Center, Los Angeles, California
  - Cedars Sinai Medical Center, Division of Pulmonary and Critical Care Medicine, Los Angeles, California
  - University of California Davis Health System, Sacramento, California
  - University of Miami, Miami, Florida
  - DBC Research Corp, Pembroke Pines, Tamarac, Florida
  - Cleveland Clinic Florida - Weston, Weston, Florida
  - University of Chicago Medical Center, Chicago, Illinois
  - LaPorte County Institute for Clinical Research, Inc., Michigan City, Indiana
  - Pulmonary Critical Care Associates of Baltimore, Towson, Maryland
  - Hannibal Clinic, Hannibal, Missouri
  - Southeastern Research Center LLC, Winston-Salem, North Carolina
  - Dayton Respiratory Research Center, Dayton, Ohio
  - Temple University School of Medicine, Philadelphia, Pennsylvania
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Renovatio Clinical-Respiratory & Sleep Disorders Specialists, The Woodlands, Texas
  - University of Texas Health Science Center at Tyler, Tyler, Texas
- LHSC - Victoria Hospital, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 21 centers in the United States and 1 center in Canada between 08 Mar 2016 (first participant first visit) and 29 Jul 2020 (last participant last visit).
Pre-assignment Details: A total of 34 participants were randomized and received the study treatment.
Groups:
- Cohort I: GLASSIA (High-end): Participants received weekly intravenous (IV) infusions of GLASSIA (lot with particle loads representing the high end within the normal range) at 60 milligrams per kilogram (mg/kg) body weight (BW) active Alpha1-Proteinase Inhibitor (A1PI) protein at a rate of 0.2 milliliters per kilogram per minute (ml/kg/min) for 25 weeks (25 planned infusions).
- Cohort II: GLASSIA (Low-end): Participants received weekly IV infusions of GLASSIA (lot with particle loads representing the low end within the normal range) at 60 mg/kg BW active A1PI protein at a rate of 0.2 ml/kg/min for 25 weeks (25 planned infusions).
Period: Overall Study
Arm/Group | Cohort I: GLASSIA (High-end) | Cohort II: GLASSIA (Low-end)
Started | 18 | 16
Completed | 17 | 14
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set consisted of all enrolled participants who received any amount of investigational product (IP), regardless of protocol deviations or non-adherence to study procedures.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort I: GLASSIA (High-end) | Cohort II: GLASSIA (Low-end) | Total
Number analyzed (Participants) | 18 | 16 | 34
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.9 (8.95) | 58.9 (9.32) | 58.4 (9.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 10 | 10 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 17 | 14 | 31
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 18 | 16 | 34
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) Potentially Related to Presence of Particle Load in the GLASSIA Solution
Description: An Adverse Events (AEs) was defined as any untoward medical occurrence in a participant administered an IP that does not necessarily have a causal relationship with the treatment. Any AE that occurs on or after the first dose of IP infusion will be considered a TEAE. A TEAE that is considered potentially related to the presence of protein aggregates (particle load) in the GLASSIA solution is defined as any embolic or thrombotic event. Number of participants with TEAEs potentially related to the presence of protein aggregates (particle load) in the GLASSIA solution were reported.
Time Frame: From start of study treatment up to Week 26
Population: Safety analysis set consisted of all enrolled participants who received any amount of IP, regardless of protocol deviations or non-adherence to study procedures.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort I: GLASSIA (High-end) | Cohort II: GLASSIA (Low-end)
Number analyzed (Participants) | 18 | 16
Participants | 0 | 0

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Reactions (ARs) Plus Suspected Adverse Reactions (ARs) Within 24 Hours Following the End of IP Infusion
Description: An Treatment-emergent AR and suspected AR was any TEAE which met any of the following criteria: a; A TEAE that began during infusion or within 24 hours (or 1 day where time of onset is not available) following the end of IP infusion, or b; A TEAE considered by either the investigator and/or the sponsor to be possibly or probably related to IP administration, or c; A TEAE for which causality assessment was missing or indeterminate. Number of participants with both treatment-emergent ARs plus suspected ARs were collectively reported.
Time Frame: From start of study treatment up to 24 hours post infusion
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort I: GLASSIA (High-end) | Cohort II: GLASSIA (Low-end)
Number analyzed (Participants) | 18 | 16
Participants | 7 | 3

3. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Reactions (ARs) Plus Suspected Adverse Reactions (ARs) Within 72 Hours Following the End of IP Infusion
Description: An Treatment-emergent AR and suspected AR was any TEAE which met any of the following criteria: a; A TEAE that began during infusion or within 72 hours (or 3 days where time of onset is not available) following the end of IP infusion, or b; A TEAE considered by either the investigator and/or the sponsor to be possibly or probably related to IP administration, or c; A TEAE for which causality assessment was missing or indeterminate. Number of participants with both treatment-emergent ARs plus suspected ARs were collectively reported.
Time Frame: From start of study treatment up to 72 hours post infusion
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort I: GLASSIA (High-end) | Cohort II: GLASSIA (Low-end)
Number analyzed (Participants) | 18 | 16
Participants | 10 | 7

4. Primary Outcome: Number of Infusions Discontinued, Slowed, or Interrupted Due to TEAEs
Description: An AE was defined as any untoward medical occurrence in a participant administered an IP that does not necessarily have a causal relationship with the treatment. Infusions may be interrupted or discontinued in an individual participant in the event of intolerable moderate to severe infusion-related AEs and/or at the discretion of the investigator. Number of infusions that are discontinued, slowed, or interrupted due to TEAEs were reported.
Time Frame: From start of study treatment up to Week 26
Population: as for outcome 1
Measure: Number; unit: Number of Infusions
Arm/Group | Cohort I: GLASSIA (High-end) | Cohort II: GLASSIA (Low-end)
Number analyzed (Participants) | 18 | 16
Number of Infusions
  Number of Infusions Discontinued due to TEAEs | 0 | 0
  Number of Infusions Slowed due to TEAEs | 1 | 0
  Number of Infusions Interrupted due to TEAEs | 0 | 0

5. Primary Outcome: Number of Participants Who Developed Binding and/or Neutralizing Anti- Alpha1-Proteinase Inhibitor(A1PI) Antibodies
Description: Development of Binding/Neutralizing Anti-A1PI Antibodies=Negative or missing at Baseline and confirmed positive at any post-infusion time point. Participants that had a positive result at Baseline and missing at all post-infusion time points were included as "No Development". Neutralizing anti-A1PI antibodies were only assessed in case of positive binding anti-A1PI antibodies. Anti-A1PI antibodies was detected using validated binding and neutralizing anti-A1PI antibody assays at a qualified immunoassay laboratory. Number of participants who developed binding and/or neutralizing anti-A1PI antibodies were reported.
Time Frame: From start of study treatment up to Week 26
Population: Safety analysis set consisted of all enrolled participants who received any amount of IP, regardless of protocol deviations or non-adherence to study procedures. Here, number analyzed signifies participants who were evaluable for this outcome measure at specific category.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort I: GLASSIA (High-end) | Cohort II: GLASSIA (Low-end)
Number analyzed (Participants) | 18 | 16
Participants
  Number of participants with binding Anti-A1PI antibodies | 1 | 1
  Number of participants with neutralizing Anti-A1PI antibodies: number analyzed (Participants) | 2 | 1
  Number of participants with neutralizing Anti-A1PI antibodies | 1 | 1

6. Primary Outcome: Change From Baseline in Antigenic Alpha1-Proteinase Inhibitor (A1PI) Levels in Epithelial Lining Fluid (ELF)
Description: Change from baseline in antigenic A1PI levels in ELF up to Week 14 was reported. Bronchoalveolar Lavage (BAL) procedures were performed at baseline and on-treatment BAL visit during GLASSIA augmentation therapy. Data for this outcome measure was analyzed and planned to be reported based on overall arm (Arms/Groups were combined as pre-specified in the study protocol).
Time Frame: Baseline up to Week 14
Population: BAL analysis set included a subset of the full analysis set (FAS). FAS included all enrolled participants who received at least 1 IP infusion and have at least 1 available antigenic or functional A1PI measurement (either from plasma or from ELF) during the treatment period.
Measure: Median (Full Range); unit: Micromolar (mcM)
Groups:
- All GLASSIA 60 mg/kg/Week: All participants who received weekly IV infusions of GLASSIA (lot with particle loads representing the High and low end within the normal range) at 60 mg/kg BW active A1PI protein at a rate of 0.2 ml/kg/min for 25 weeks (25 planned infusions).
Arm/Group | All GLASSIA 60 mg/kg/Week
Number analyzed (Participants) | 16
Micromolar (mcM) | 0.515 [0.08 to 2.41]
Statistical Analysis 1: Comparison: All GLASSIA 60 mg/kg/Week; Statistical analysis was collected and assessed based on A1P1 Levels at baseline and On-treatment BAL visit; Test type: Other; p < 0.001, Mixed-effects model; Geometric Mean Ratio = 5.398

7. Primary Outcome: Change From Baseline in Functional Alpha1-Proteinase Inhibitor(A1PI) Levels in Epithelial Lining Fluid (ELF)
Description: Change from baseline in functional A1PI (also known as Anti-Neutrophil Elastase Capacity [ANEC]) levels in ELF up to Week 14 was reported. BAL procedures were performed at baseline and on-treatment BAL visit during GLASSIA augmentation therapy. Data for this outcome measure was analyzed and planned to be reported based on overall arm (Arms/Groups were combined as pre-specified in the study protocol).
Time Frame: Baseline up to Week 14
Population: BAL analysis set included a subset of the FAS. FAS included all enrolled participants who received at least 1 IP infusion and have at least 1 available antigenic or functional A1PI measurement (either from plasma or from ELF) during the treatment period.
Measure: Median (Full Range); unit: mcM
Groups:
- All GLASSIA 60 mg/kg/Week: All participants who received weekly IV infusions of GLASSIA (lot with particle loads representing the High and low end within the normal range) at 60 mg/kg BW active A1PI protein administered at a rate of 0.2 ml/kg/min for 25 weeks (25 planned infusions).
Arm/Group | All GLASSIA 60 mg/kg/Week
Number analyzed (Participants) | 16
mcM | 0.256 [-0.28 to 1.54]
Statistical Analysis 1: Comparison: All GLASSIA 60 mg/kg/Week; Statistical analysis was collected and assessed based on functional A1P1 Levels at baseline and On-treatment BAL visit; Test type: Other; p < 0.001, mixed-effects model; Geometric Mean Ratio = 2.259

8. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An AEs was defined as any untoward medical occurrence in a participant administered an IP that does not necessarily have a causal relationship with the treatment. Any AE that occurs on or after the first dose of IP infusion will be considered a TEAE.
Time Frame: From start of study treatment up to Week 26
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort I: GLASSIA (High-end) | Cohort II: GLASSIA (Low-end)
Number analyzed (Participants) | 18 | 16
Participants | 13 | 9

9. Secondary Outcome: Number of Participants Who Experienced a Shift From Normal or Clinically Non-significant Abnormal Laboratory Values at Baseline to Clinically Significant Abnormal Laboratory Values at Week 13, 25, and 26
Description: Clinical laboratory values included Hematology (hemoglobin, leukocytes, neutrophils, reticulocytes/erythrocytes [Ret/Ery], platelets); Chemistry (sodium, potassium, albumin, alanine aminotransferase [AA], aspartate aminotransferase [ASA], alkaline phosphatase [AP], lactate dehydrogenase [LD], gamma glutamyl transferase [GGT], bilirubin, direct bilirubin [DB], creatinine, creatine kinase [CK], glucose); Urinalysis (erythrocytes urine [EU], protein urine [PU], specific gravity [SG], pH) and Immunology (Complement C3, Complement C4). Assessment if a value was normal, clinically non-significant abnormal, or clinically significant abnormal was done by the investigator. Number of participants who experienced a shift from normal or clinically non-significant (NCS) abnormal laboratory values at baseline [BL] to clinically significant (CS) abnormal laboratory values at Week 13, 25 and 26 were reported.
Time Frame: Baseline, Week 13, 25 and 26
Population: Safety analysis set consisted of all enrolled participants who received any amount of IP, regardless of protocol deviations or non-adherence to study procedures. Here, number of participants analyzed signifies participants who were evaluable for this outcome measure and number analyzed signifies participants who were evaluable for at specific time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort I: GLASSIA (High-end) | Cohort II: GLASSIA (Low-end)
Number analyzed (Participants) | 17 | 15
Participants
  Hemoglobin: Normal at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 14 | 14
  Hemoglobin: Normal at BL→Abnormal-CS at Week 13 | 0 | 0
  Hemoglobin: Abnormal-NCS at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 14 | 14
  Hemoglobin: Abnormal-NCS at BL→Abnormal-CS at Week 13 | 0 | 0
  Hemoglobin: Normal at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 16 | 14
  Hemoglobin: Normal at BL→Abnormal-CS at Week 25 | 0 | 0
  Hemoglobin: Abnormal-NCS at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 16 | 14
  Hemoglobin: Abnormal-NCS at BL→Abnormal-CS at Week 25 | 0 | 0
  Hemoglobin: Normal at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 17 | 12
  Hemoglobin: Normal at BL→Abnormal-CS at Week 26 | 0 | 0
  Hemoglobin: Abnormal-NCS at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 17 | 12
  Hemoglobin: Abnormal-NCS at BL→Abnormal-CS at Week 26 | 0 | 0
  Leukocytes: Normal at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 13 | 14
  Leukocytes: Normal at BL→Abnormal-CS at Week 13 | 0 | 0
  Leukocytes: Abnormal-NCS at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 13 | 14
  Leukocytes: Abnormal-NCS at BL→Abnormal-CS at Week 13 | 0 | 0
  Leukocytes: Normal at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 16 | 14
  Leukocytes: Normal at BL→Abnormal-CS at Week 25 | 0 | 0
  Leukocytes: Abnormal-NCS at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 16 | 14
  Leukocytes: Abnormal-NCS at BL→Abnormal-CS at Week 25 | 0 | 0
  Leukocytes: Normal at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 17 | 12
  Leukocytes: Normal at BL→Abnormal-CS at Week 26 | 0 | 0
  Leukocytes: Abnormal-NCS at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 17 | 12
  Leukocytes: Abnormal-NCS at BL→Abnormal-CS at Week 26 | 0 | 0
  Neutrophils: Normal at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 13 | 14
  Neutrophils: Normal at BL→Abnormal-CS at Week 13 | 0 | 0
  Neutrophils: Abnormal-NCS at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 13 | 14
  Neutrophils: Abnormal-NCS at BL→Abnormal-CS at Week 13 | 0 | 0
  Neutrophils: Normal at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 16 | 14
  Neutrophils: Normal at BL→Abnormal-CS at Week 25 | 1 | 0
  Neutrophils: Abnormal-NCS at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 16 | 14
  Neutrophils: Abnormal-NCS at BL→Abnormal-CS at Week 25 | 0 | 0
  Neutrophils: Normal at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 17 | 12
  Neutrophils: Normal at BL→Abnormal-CS at Week 26 | 0 | 0
  Neutrophils: Abnormal-NCS at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 17 | 12
  Neutrophils: Abnormal-NCS at BL→Abnormal-CS at Week 26 | 0 | 0
  Ret/Ery: Normal at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 14 | 14
  Ret/Ery: Normal at BL→Abnormal-CS at Week 13 | 1 | 0
  Ret/Ery: Abnormal-NCS at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 14 | 14
  Ret/Ery: Abnormal-NCS at BL→Abnormal-CS at Week 13 | 0 | 0
  Ret/Ery: Normal at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 16 | 14
  Ret/Ery: Normal at BL→Abnormal-CS at Week 25 | 0 | 0
  Ret/Ery: Abnormal-NCS at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 16 | 14
  Ret/Ery: Abnormal-NCS at BL→Abnormal-CS at Week 25 | 0 | 0
  Ret/Ery: Normal at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 17 | 12
  Ret/Ery: Normal at BL→Abnormal-CS at Week 26 | 1 | 0
  Ret/Ery: Abnormal-NCS at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 17 | 12
  Ret/Ery: Abnormal-NCS at BL→Abnormal-CS at Week 26 | 0 | 0
  Platelets: Normal at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 13 | 14
  Platelets: Normal at BL→Abnormal-CS at Week 13 | 0 | 0
  Platelets: Abnormal-NCS at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 13 | 14
  Platelets: Abnormal-NCS at BL→Abnormal-CS at Week 13 | 0 | 0
  Platelets: Normal at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 15 | 14
  Platelets: Normal at BL→Abnormal-CS at Week 25 | 0 | 0
  Platelets: Abnormal-NCS at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 15 | 14
  Platelets: Abnormal-NCS at BL→Abnormal-CS at Week 25 | 0 | 0
  Platelets: Normal at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 16 | 12
  Platelets: Normal at BL→Abnormal-CS at Week 26 | 0 | 0
  Platelets: Abnormal-NCS at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 16 | 12
  Platelets: Abnormal-NCS at BL→Abnormal-CS at Week 26 | 0 | 0
  Sodium: Normal at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 13 | 13
  Sodium: Normal at BL→Abnormal-CS at Week 13 | 0 | 0
  Sodium: Abnormal-NCS at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 13 | 13
  Sodium: Abnormal-NCS at BL→Abnormal-CS at Week 13 | 0 | 0
  Sodium: Normal at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 15 | 14
  Sodium: Normal at BL→Abnormal-CS at Week 25 | 0 | 0
  Sodium: Abnormal-NCS at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 15 | 14
  Sodium: Abnormal-NCS at BL→Abnormal-CS at Week 25 | 0 | 0
  Sodium: Normal at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 17 | 13
  Sodium: Normal at BL→Abnormal-CS at Week 26 | 0 | 0
  Sodium: Abnormal-NCS at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 17 | 13
  Sodium: Abnormal-NCS at BL→Abnormal-CS at Week 26 | 0 | 0
  Potassium: Normal at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 13 | 13
  Potassium: Normal at BL→Abnormal-CS at Week 13 | 0 | 0
  Potassium: Abnormal-NCS at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 13 | 13
  Potassium: Abnormal-NCS at BL→Abnormal-CS at Week 13 | 0 | 0
  Potassium: Normal at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 15 | 14
  Potassium: Normal at BL→Abnormal-CS at Week 25 | 0 | 0
  Potassium: Abnormal-NCS at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 15 | 14
  Potassium: Abnormal-NCS at BL→Abnormal-CS at Week 25 | 0 | 0
  Potassium: Normal at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 17 | 13
  Potassium: Normal at BL→Abnormal-CS at Week 26 | 0 | 0
  Potassium: Abnormal-NCS at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 17 | 13
  Potassium: Abnormal-NCS at BL→Abnormal-CS at Week 26 | 0 | 0
  Albumin: Normal at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 13 | 13
  Albumin: Normal at BL→Abnormal-CS at Week 13 | 0 | 0
  Albumin: Abnormal-NCS at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 13 | 13
  Albumin: Abnormal-NCS at BL→Abnormal-CS at Week 13 | 0 | 0
  Albumin: Normal at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 15 | 14
  Albumin: Normal at BL→Abnormal-CS at Week 25 | 0 | 0
  Albumin: Abnormal-NCS at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 15 | 14
  Albumin: Abnormal-NCS at BL→Abnormal-CS at Week 25 | 0 | 0
  Albumin: Normal at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 17 | 13
  Albumin: Normal at BL→Abnormal-CS at Week 26 | 0 | 0
  Albumin: Abnormal-NCS at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 17 | 13
  Albumin: Abnormal-NCS at BL→Abnormal-CS at Week 26 | 0 | 0
  AA: Normal at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 13 | 13
  AA: Normal at BL→Abnormal-CS at Week 13 | 0 | 0
  AA: Abnormal-NCS at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 13 | 13
  AA: Abnormal-NCS at BL→Abnormal-CS at Week 13 | 0 | 0
  AA: Normal at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 15 | 14
  AA: Normal at BL→Abnormal-CS at Week 25 | 0 | 0
  AA: Abnormal-NCS at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 15 | 14
  AA: Abnormal-NCS at BL→Abnormal-CS at Week 25 | 0 | 0
  AA: Normal at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 17 | 13
  AA: Normal at BL→Abnormal-CS at Week 26 | 0 | 0
  AA: Abnormal-NCS at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 17 | 13
  AA: Abnormal-NCS at BL→Abnormal-CS at Week 26 | 0 | 0
  ASA: Normal at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 13 | 13
  ASA: Normal at BL→Abnormal-CS at Week 13 | 0 | 0
  ASA: Abnormal-NCS at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 13 | 13
  ASA: Abnormal-NCS at BL→Abnormal-CS at Week 13 | 0 | 0
  ASA: Normal at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 14 | 14
  ASA: Normal at BL→Abnormal-CS at Week 25 | 0 | 0
  ASA: Abnormal-NCS at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 14 | 14
  ASA: Abnormal-NCS at BL→Abnormal-CS at Week 25 | 0 | 0
  ASA: Normal at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 17 | 13
  ASA: Normal at BL→Abnormal-CS at Week 26 | 0 | 0
  ASA: Abnormal-NCS at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 17 | 13
  ASA: Abnormal-NCS at BL→Abnormal-CS at Week 26 | 0 | 0
  AP: Normal at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 13 | 13
  AP: Normal at BL→Abnormal-CS at Week 13 | 0 | 0
  AP: Abnormal-NCS at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 13 | 13
  AP: Abnormal-NCS at BL→Abnormal-CS at Week 13 | 0 | 0
  AP: Normal at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 15 | 14
  AP: Normal at BL→Abnormal-CS at Week 25 | 0 | 0
  AP: Abnormal-NCS at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 15 | 14
  AP: Abnormal-NCS at BL→Abnormal-CS at Week 25 | 0 | 0
  AP: Normal at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 17 | 13
  AP: Normal at BL→Abnormal-CS at Week 26 | 0 | 0
  AP: Abnormal-NCS at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 17 | 13
  AP: Abnormal-NCS at BL→Abnormal-CS at Week 26 | 0 | 0
  LD: Normal at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 13 | 13
  LD: Normal at BL→Abnormal-CS at Week 13 | 0 | 0
  LD: Abnormal-NCS at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 13 | 13
  LD: Abnormal-NCS at BL→Abnormal-CS at Week 13 | 0 | 0
  LD: Normal at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 14 | 14
  LD: Normal at BL→Abnormal-CS at Week 25 | 0 | 0
  LD: Abnormal-NCS at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 14 | 14
  LD: Abnormal-NCS at BL→Abnormal-CS at Week 25 | 0 | 0
  LD: Normal at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 17 | 13
  LD: Normal at BL→Abnormal-CS at Week 26 | 0 | 0
  LD: Abnormal-NCS at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 17 | 13
  LD: Abnormal-NCS at BL→Abnormal-CS at Week 26 | 0 | 0
  GGT: Normal at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 13 | 13
  GGT: Normal at BL→Abnormal-CS at Week 13 | 0 | 0
  GGT: Abnormal-NCS at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 13 | 13
  GGT: Abnormal-NCS at BL→Abnormal-CS at Week 13 | 0 | 0
  GGT: Normal at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 15 | 14
  GGT: Normal at BL→Abnormal-CS at Week 25 | 0 | 0
  GGT: Abnormal-NCS at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 15 | 14
  GGT: Abnormal-NCS at BL→Abnormal-CS at Week 25 | 0 | 0
  GGT: Normal at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 17 | 13
  GGT: Normal at BL→Abnormal-CS at Week 26 | 0 | 0
  GGT: Abnormal-NCS at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 17 | 13
  GGT: Abnormal-NCS at BL→Abnormal-CS at Week 26 | 0 | 0
  Bilirubin: Normal at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 13 | 13
  Bilirubin: Normal at BL→Abnormal-CS at Week 13 | 0 | 0
  Bilirubin: Abnormal-NCS at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 13 | 13
  Bilirubin: Abnormal-NCS at BL→Abnormal-CS at Week 13 | 0 | 0
  Bilirubin: Normal at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 15 | 14
  Bilirubin: Normal at BL→Abnormal-CS at Week 25 | 0 | 0
  Bilirubin: Abnormal-NCS at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 15 | 14
  Bilirubin: Abnormal-NCS at BL→Abnormal-CS at Week 25 | 0 | 0
  Bilirubin: Normal at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 17 | 13
  Bilirubin: Normal at BL→Abnormal-CS at Week 26 | 0 | 0
  Bilirubin: Abnormal-NCS at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 17 | 13
  Bilirubin: Abnormal-NCS at BL→Abnormal-CS at Week 26 | 0 | 0
  DB: Normal at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 13 | 13
  DB: Normal at BL→Abnormal-CS at Week 13 | 0 | 0
  DB: Abnormal-NCS at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 13 | 13
  DB: Abnormal-NCS at BL→Abnormal-CS at Week 13 | 0 | 0
  DB: Normal at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 14 | 14
  DB: Normal at BL→Abnormal-CS at Week 25 | 0 | 0
  DB: Abnormal-NCS at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 14 | 14
  DB: Abnormal-NCS at BL→Abnormal-CS at Week 25 | 0 | 0
  DB: Normal at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 17 | 13
  DB: Normal at BL→Abnormal-CS at Week 26 | 0 | 0
  DB: Abnormal-NCS at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 17 | 13
  DB: Abnormal-NCS at BL→Abnormal-CS at Week 26 | 0 | 0
  Creatinine: Normal at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 13 | 13
  Creatinine: Normal at BL→Abnormal-CS at Week 13 | 0 | 0
  Creatinine: Abnormal-NCS at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 13 | 13
  Creatinine: Abnormal-NCS at BL→Abnormal-CS at Week 13 | 0 | 0
  Creatinine: Normal at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 15 | 14
  Creatinine: Normal at BL→Abnormal-CS at Week 25 | 0 | 0
  Creatinine: Abnormal-NCS at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 15 | 14
  Creatinine: Abnormal-NCS at BL→Abnormal-CS at Week 25 | 0 | 0
  Creatinine: Normal at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 17 | 13
  Creatinine: Normal at BL→Abnormal-CS at Week 26 | 0 | 0
  Creatinine: Abnormal-NCS at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 17 | 13
  Creatinine: Abnormal-NCS at BL→Abnormal-CS at Week 26 | 0 | 0
  CK: Normal at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 13 | 13
  CK: Normal at BL→Abnormal-CS at Week 13 | 0 | 0
  CK: Abnormal-NCS at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 13 | 13
  CK: Abnormal-NCS at BL→Abnormal-CS at Week 13 | 0 | 0
  CK: Normal at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 15 | 14
  CK: Normal at BL→Abnormal-CS at Week 25 | 1 | 0
  CK: Abnormal-NCS at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 15 | 14
  CK: Abnormal-NCS at BL→Abnormal-CS at Week 25 | 0 | 0
  CK: Normal at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 17 | 13
  CK: Normal at BL→Abnormal-CS at Week 26 | 0 | 0
  CK: Abnormal-NCS at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 17 | 13
  CK: Abnormal-NCS at BL→Abnormal-CS at Week 26 | 0 | 0
  Glucose: Normal at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 13 | 13
  Glucose: Normal at BL→Abnormal-CS at Week 13 | 0 | 0
  Glucose: Abnormal-NCS at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 13 | 13
  Glucose: Abnormal-NCS at BL→Abnormal-CS at Week 13 | 0 | 0
  Glucose: Normal at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 15 | 14
  Glucose: Normal at BL→Abnormal-CS at Week 25 | 0 | 0
  Glucose: Abnormal-NCS at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 15 | 14
  Glucose: Abnormal-NCS at BL→Abnormal-CS at Week 25 | 0 | 0
  Glucose: Normal at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 17 | 13
  Glucose: Normal at BL→Abnormal-CS at Week 26 | 0 | 0
  Glucose: Abnormal-NCS at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 17 | 13
  Glucose: Abnormal-NCS at BL→Abnormal-CS at Week 26 | 0 | 0
  EU: Normal at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 1 | 1
  EU: Normal at BL→Abnormal-CS at Week 13 | 0 | 0
  EU: Abnormal-NCS at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 1 | 1
  EU: Abnormal-NCS at BL→Abnormal-CS at Week 13 | 0 | 0
  EU: Normal at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 0 | 0
  EU: Abnormal-NCS at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 0 | 0
  EU: Normal at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 1 | 0
  EU: Normal at BL→Abnormal-CS at Week 26 | 0 | 0
  EU: Abnormal-NCS at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 1 | 0
  EU: Abnormal-NCS at BL→Abnormal-CS at Week 26 | 0 | 0
  PU: Normal at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 14 | 14
  PU: Normal at BL→Abnormal-CS at Week 13 | 0 | 0
  PU: Abnormal-NCS at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 14 | 14
  PU: Abnormal-NCS at BL→Abnormal-CS at Week 13 | 0 | 0
  PU: Normal at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 16 | 15
  PU: Normal at BL→Abnormal-CS at Week 25 | 0 | 0
  PU: Abnormal-NCS at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 16 | 15
  PU: Abnormal-NCS at BL→Abnormal-CS at Week 25 | 0 | 0
  PU: Normal at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 16 | 13
  PU: Normal at BL→Abnormal-CS at Week 26 | 0 | 0
  PU: Abnormal-NCS at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 16 | 13
  PU: Abnormal-NCS at BL→Abnormal-CS at Week 26 | 0 | 0
  SG: Normal at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 14 | 14
  SG: Normal at BL→Abnormal-CS at Week 13 | 0 | 0
  SG: Abnormal-NCS at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 14 | 14
  SG: Abnormal-NCS at BL→Abnormal-CS at Week 13 | 0 | 0
  SG: Normal at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 16 | 15
  SG: Normal at BL→Abnormal-CS at Week 25 | 0 | 0
  SG: Abnormal-NCS at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 16 | 15
  SG: Abnormal-NCS at BL→Abnormal-CS at Week 25 | 0 | 0
  SG: Normal at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 16 | 13
  SG: Normal at BL→Abnormal-CS at Week 26 | 0 | 0
  SG: Abnormal-NCS at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 16 | 13
  SG: Abnormal-NCS at BL→Abnormal-CS at Week 26 | 0 | 0
  pH: Normal at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 14 | 14
  pH: Normal at BL→Abnormal-CS at Week 13 | 0 | 0
  pH: Abnormal-NCS at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 14 | 14
  pH: Abnormal-NCS at BL→Abnormal-CS at Week 13 | 0 | 0
  pH: Normal at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 16 | 15
  pH: Normal at BL→Abnormal-CS at Week 25 | 0 | 0
  pH: Abnormal-NCS at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 16 | 15
  pH: Abnormal-NCS at BL→Abnormal-CS at Week 25 | 0 | 0
  pH: Normal at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 16 | 13
  pH: Normal at BL→Abnormal-CS at Week 26 | 0 | 0
  pH: Abnormal-NCS at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 16 | 13
  pH: Abnormal-NCS at BL→Abnormal-CS at Week 26 | 0 | 0
  C3: Normal at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 12 | 14
  C3: Normal at BL→Abnormal-CS at Week 13 | 0 | 0
  C3: Abnormal-NCS at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 12 | 14
  C3: Abnormal-NCS at BL→Abnormal-CS at Week 13 | 0 | 0
  C3: Normal at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 14 | 15
  C3: Normal at BL→Abnormal-CS at Week 25 | 0 | 0
  C3: Abnormal-NCS at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 14 | 15
  C3: Abnormal-NCS at BL→Abnormal-CS at Week 25 | 0 | 0
  C3: Normal at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 16 | 13
  C3: Normal at BL→Abnormal-CS at Week 26 | 0 | 0
  C3: Abnormal-NCS at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 16 | 13
  C3: Abnormal-NCS at BL→Abnormal-CS at Week 26 | 0 | 0
  C4: Normal at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 12 | 14
  C4: Normal at BL→Abnormal-CS at Week 13 | 0 | 0
  C4: Abnormal-NCS at BL→Abnormal-CS at Week 13: number analyzed (Participants) | 12 | 14
  C4: Abnormal-NCS at BL→Abnormal-CS at Week 13 | 0 | 0
  C4: Normal at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 14 | 15
  C4: Normal at BL→Abnormal-CS at Week 25 | 0 | 0
  C4: Abnormal-NCS at BL→Abnormal-CS at Week 25: number analyzed (Participants) | 14 | 15
  C4: Abnormal-NCS at BL→Abnormal-CS at Week 25 | 0 | 0
  C4: Normal at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 16 | 13
  C4: Normal at BL→Abnormal-CS at Week 26 | 0 | 0
  C4: Abnormal-NCS at BL→Abnormal-CS at Week 26: number analyzed (Participants) | 16 | 13
  C4: Abnormal-NCS at BL→Abnormal-CS at Week 26 | 0 | 0

10. Secondary Outcome: Number of Participants With Treatment-Emergent Seroconversion or Positive Nucleic Acid Test (NAT) for Parvovirus B19 (B19V)
Description: Viral testing for B19V consisted of viral serology or NAT for B19V (Parvovirus B19 IgG Antibody, Parvovirus B19 IgM Antibody, Parvovirus B19 DNA Quant real-time polymerase chain reaction [RT-PCR]). Number of participants with treatment-emergent seroconversion or positive NAT for B19V were reported.
Time Frame: From start of study treatment up to Week 26
Population: Safety analysis set consisted of all enrolled participants who received any amount of IP, regardless of protocol deviations or non-adherence to study procedures. Here, "number analyzed" signifies those participants who were evaluable for this outcome measure at specific category.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort I: GLASSIA (High-end) | Cohort II: GLASSIA (Low-end)
Number analyzed (Participants) | 18 | 16
Participants
  Number of participants with parvovirus B19 IgG antibody | 0 | 1
  Number of participants with parvovirus B19 IgM antibody: number analyzed (Participants) | 18 | 15
  Number of participants with parvovirus B19 IgM antibody | 0 | 0
  Number of participants with Parvovirus B19 DNA Quant RT-PCR: number analyzed (Participants) | 18 | 15
  Number of participants with Parvovirus B19 DNA Quant RT-PCR | 0 | 0

ADVERSE EVENTS:
Time Frame: From start of study treatment up to Week 26
Groups:
- GLASSIA (High-end): Participants received weekly intravenous (IV) infusions of GLASSIA (lot with particle loads representing the high end within) at 60 milligrams per kilogram (mg/kg) body weight (BW) active A1PI protein at a rate of 0.2 milliliters per kilogram per minute (ml/kg/min) for 25 weeks (25 planned infusions).
- GLASSIA (Low-end): Participants received weekly IV infusions of GLASSIA (lot with particle loads representing the low end within the normal range) at 60 mg/kg BW active A1PI protein at a rate of 0.2 ml/kg/min for 25 weeks (25 planned infusions).
Arm/Group | GLASSIA (High-end) | GLASSIA (Low-end)
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/16
Serious Adverse Events (participants affected / at risk) | 1/18 | 1/16
Other Adverse Events (participants affected / at risk) | 13/18 | 9/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GLASSIA (High-end) (N=18) | GLASSIA (Low-end) (N=16)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GLASSIA (High-end) (N=18) | GLASSIA (Low-end) (N=16)
Eye irritation (Eye disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Lip dry (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Body tinea (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1)
Ear infection (Infections and infestations) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (6) | 1 (2)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (4)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 1 (1)
Blood bicarbonate decreased (Investigations) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Oxygen saturation decreased (Investigations) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (2)
Lethargy (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Urine abnormality (Renal and urinary disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (8):
  • Study Protocol: Amendment 7 (2020-05-26): https://cdn.clinicaltrials.gov/large-docs/61/NCT02525861/Prot_000.pdf
  • Study Protocol: Amendment 1 (2015-01-19): https://cdn.clinicaltrials.gov/large-docs/61/NCT02525861/Prot_001.pdf
  • Study Protocol: Amendment 2 (2015-05-07): https://cdn.clinicaltrials.gov/large-docs/61/NCT02525861/Prot_002.pdf
  • Study Protocol: Amendment 4 (2016-01-15): https://cdn.clinicaltrials.gov/large-docs/61/NCT02525861/Prot_003.pdf
  • Study Protocol: Amendment 5 (2017-11-21): https://cdn.clinicaltrials.gov/large-docs/61/NCT02525861/Prot_004.pdf
  • Study Protocol: Amendment 6 (2018-08-27): https://cdn.clinicaltrials.gov/large-docs/61/NCT02525861/Prot_005.pdf
  • Study Protocol: Amendment 3 (2015-08-26): https://cdn.clinicaltrials.gov/large-docs/61/NCT02525861/Prot_006.pdf
  • Statistical Analysis Plan (2020-09-09): https://cdn.clinicaltrials.gov/large-docs/61/NCT02525861/SAP_007.pdf